CLINICAL TRIAL: NCT02407223
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Ustekinumab in the Treatment of Subjects With Active Nonradiographic Axial Spondyloarthritis
Brief Title: An Efficacy and Safety Study of Ustekinumab in Participants With Active Nonradiographic Axial Spondyloarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped because ustekinumab did not achieve key endpoints in a related study. The safety profile was consistent with past ustekinumab studies.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106995; CNTO1275AKS3003 (Other: Janssen Research & Development, LLC); 2015-000289-67 (EudraCT Number)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Nonradiographic Axial Spondylitis, Ankylosing
Keywords: Nonradiographic Axial Spondylitis, Ankylosing; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Device: No

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo subcutaneously (SC) at Weeks 0, 4, 16, and 20. At Week 24, all participants (except those who early escaped) will crossover to receive ustekinumab 45 or 90 milligram (mg) SC at Weeks 24 and 28 followed by every 12 weeks up to Week 52. At Week 16, participants in placebo group with < 10% improvement from baseline in both total back pain and morning stiffness measures at Week 12 and 16 will enter early escape to receive ustekinumab 45 mg or 90 mg at Weeks 16, 20, and 28 followed by every 12 weeks up to Week 52. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and 52 will be re-randomized to receive placebo or ustekinumab every 12 weeks up to Week 88. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or 52 will continue with ustekinumab every 12 weeks up to Week 88. NOTE: Intervention Description should have no more than 800 characters.
  Interventions: Drug: Group 1: Placebo
- Group 2: Ustekinumab 45 milligram (mg) (Experimental): Participants will receive ustekinumab 45 mg subcutaneously at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants will receive placebo subcutaneously to maintain the blind. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and Week 52 will be re-randomized to receive either placebo or ustekinumab 45 mg every 12 weeks in a blinded fashion. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or Week 52 will continue receiving ustekinumab 45 mg every 12 weeks through Week 88.
  Interventions: Drug: Group 2: Ustekinumab 45 mg
- Group 3: Ustekinumab 90 mg (Experimental): Participants will receive ustekinumab 90 mg subcutaneously at Weeks 0 and 4, followed by every four weeks through Week 52. At Weeks 20 and 24, participants will receive placebo subcutaneously to maintain the blind. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and Week 52 will receive either placebo or ustekinumab 90 mg every 12 weeks in a blinded fashion. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or Week 52 will continue receiving ustekinumab 90 mg every 12 weeks through Week 88.
  Interventions: Drug: Group 3: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Group 1: Placebo — Participants will receive placebo SC at Weeks 0, 4, 16, and 20. At Week 24, all participants (except those who early escaped) will crossover to receive ustekinumab 45 or 90 mg SC at Weeks 24 and 28 followed by every 12 weeks up to Week 52. At Week 16, participants in placebo group with < 10% improvement from baseline in both total back pain and morning stiffness measures at Week 12 and 16 will enter early escape to receive ustekinumab 45 mg or 90 mg at Weeks 16, 20, and 28 followed by every 12 weeks up to Week 52. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and 52 will be re-randomized to receive placebo or ustekinumab every 12 weeks up to Week 88. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or 52 will continue with ustekinumab every 12 weeks up to Week 88.
  Arms: Group 1: Placebo
Drug: Group 2: Ustekinumab 45 mg — Participants will receive ustekinumab 45 mg subcutaneously at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants will receive placebo subcutaneously to maintain the blind. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and Week 52 will be re-randomized to receive either placebo or ustekinumab 45 mg every 12 weeks in a blinded fashion. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or Week 52 will continue receiving ustekinumab 45 mg every 12 weeks through Week 88.
  Arms: Group 2: Ustekinumab 45 milligram (mg)
Drug: Group 3: Ustekinumab 90 mg — Participants will receive ustekinumab 90 mg subcutaneously at Weeks 0 and 4, followed by every four weeks through Week 52. At Weeks 20 and 24, participants will receive placebo subcutaneously to maintain the blind. At Week 52, participants who achieved inactive disease by ASDAS (ESR) <1.3 at both Week 40 and Week 52 will receive either placebo or ustekinumab 90 mg every 12 weeks in a blinded fashion. At Week 52, participants who did not achieve inactive disease by ASDAS (ESR) <1.3 at Week 40 or Week 52 will continue receiving ustekinumab 90 mg every 12 weeks through Week 88.
  Arms: Group 3: Ustekinumab 90 mg

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ustekinumab in adult participants with active nonradiographic axial spondyloarthritis (nr-AxSpA) measured by the reduction in signs and symptoms of nonradiographic axial spondyloarthritis (nr-AxSpA).

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of ustekinumab in the treatment of participants with active non-radiographic axial spondylo arthritis. Participants will receive either placebo or ustekinumab 45 or 90 milligram (mg). Participants will primarily be assessed for Assessment of Spondylo Arthritis (ASAS) International Society criteria 20 at Week 24. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be classified as having nonradiographic axial spondyloarthritis (nr-AxSpA) based on 2009 Assessment of SpondyloArthritis International Society (ASAS) criteria
* Must have an age at nr-AxSpA onset of <= 45 years
* Must have at screening or active inflammation on magnetic resonance imaging (MRI) as evidenced by the central readers and no radiographic sacroiliitis that fulfills the 1984 modified New York Criteria
* Must have symptoms of active disease at screening and at baseline, as evidenced by both a BASDAI score of >= 4 and a visual analogue scale (VAS) score for total back pain of more than or equal to (>=) 4, each on a scale of 0 to 10

Exclusion Criteria:

* Have radiographic sacroiliitis fulfilling the 1984 modified New York Criteria
* Have other inflammatory diseases that might confound the evaluations of benefit from the ustekinumab therapy
* Have received any systemic immunosuppressives or disease-modifying anti-rheumatic drug (DMARDs) other than methotrexate (MTX), sulfasalazine (SSZ), or hydroxychloroquine (HCQ) within 4 weeks prior to first administration of study agent
* Have received epidural, intra-articular, intramuscular (IM), or intravenous (IV) corticosteroids, including adrenocorticotropic hormone during the 4 weeks prior to first administration of study agent
* Have received prior biologic therapy other than anti-TNFα
* Have received more than 1 prior anti-TNFα agent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (90):
- Argentina (5):
  - Buenos Aires
  - Ciudad de Buenos Aires
  - Ciudad de La Plata
  - Ciudad de San Miguel de Tucuman
  - Córdoba
- Australia (6):
  - Geelong
  - Hobart
  - Kogarah
  - Queensland
  - Woodville South
  - Woolloongabba
- Belgium (5):
  - Genk
  - Ghent
  - Leuven
  - Liège
  - Merksem
- Czechia (8):
  - Brno
  - Bruntál
  - Kladno
  - Ostrava
  - Pardubice
  - Prague
  - Uherské Hradiště
  - Zlín
- France (6):
  - Boulogne-Billancourt
  - Chambray-lès-Tours
  - Échirolles
  - Montpellier, Herault
  - Paris
  - Toulouse
- Germany (7):
  - Bad Nauheim
  - Berlin
  - Cologne
  - Hamburg
  - Hanover
  - Herne
  - Olsberg
- Hungary (8):
  - Budapest
  - Debrecen
  - Esztergom
  - Kistarcsa
  - Nyíregyháza
  - Székesfehérvár
  - Szolnok
  - Veszprém
- Mexico (4):
  - Chihuahua City
  - Culiacán
  - Guadalajara
  - México
- Poland (5):
  - Bydgoszcz
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
- Russia (13):
  - Chelyabinsk
  - Chita
  - Kemerovo
  - Kirov
  - Moscow
  - Novosibirsk
  - Orenburg
  - Petrozavodsk
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Ulyanovsk
  - Zelenograd
- South Korea (3):
  - Gwangju
  - Incheon
  - Seoul
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (8):
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Ternopil
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (7):
  - Bath
  - Leeds
  - Leytonstone
  - London
  - Norwich
  - Staffordshire
  - Torquay

REFERENCES:
- [Derived] Deodhar A, Gensler LS, Sieper J, Clark M, Calderon C, Wang Y, Zhou Y, Leu JH, Campbell K, Sweet K, Harrison DD, Hsia EC, van der Heijde D. Three Multicenter, Randomized, Double-Blind, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Ustekinumab in Axial Spondyloarthritis. Arthritis Rheumatol. 2019 Feb;71(2):258-270. doi: 10.1002/art.40728. Epub 2018 Dec 29. PMID 30225992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 356 participants were randomized and received treatment (116 participants to placebo, 118 participants to ustekinumab 45 milligram [mg], and 122 participants to ustekinumab 90 mg).
Groups:
- Placebo: Participants received placebo subcutaneous (SC) at Week 0,4,16 and 20. At Week 16, participants in placebo group who qualified for early escape (EE) criteria (with <10 % improvement from baseline in both total back pain and morning stiffness measures at Week 12 and 16) re-randomized to receive ustekinumab 45mg or 90mg at Week 16,20,28 followed by every 12 Weeks (q12w) through Week 52. Participants received placebo SC at Week 24 to maintain blind. At Week 24, remaining participants in placebo group who did not meet EE criteria, re-randomized to receive ustekinumab 45mg or 90mg at Week 24, 28 followed by q12w through Week 52. At Week 52, participants who achieved inactive disease ASDAS [ESR]<1.3 at Week 40, 52 underwent re-randomization to either ustekinumab or placebo. Participants who did not achieve inactive disease either at Week 40 or 52 received previously assigned ustekinumab dose at scheduled visits. Last dose was scheduled for Week 88 and last study visit for Week 100.
- Ustekinumab 45mg: Participants received ustekinumab 45 mg SC at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind. At Week 52, all participants who achieved inactive disease (Ankylosing Spondylitis Disease Activity Score [ASDAS] erythrocyte sedimentation rate [ESR] less than [<] 1.3) at both Week 40 and 52 underwent re-randomization to either Ustekinumab or placebo. Participants who did not achieve inactive disease at either Week 40 or 52 received previously assigned ustekinumab dose at their scheduled visits. Last dose was scheduled for Week 88 and last study visit for Week 100.
- Ustekinumab 90mg: Participants received ustekinumab 90 mg SC at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind. At Week 52, all participants who achieved inactive disease (ASDAS ESR<1.3) at both Week 40 and 52 underwent re-randomization to either Ustekinumab or placebo. Participants who did not achieve inactive disease at either Week 40 or 52 received previously assigned ustekinumab dose at their scheduled visits. Last dose was scheduled for Week 88 and last study visit for Week 100.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Started | 116 | 118 | 122
Early Escape at Week 16 | 22 (Study discontinuation/completion reported under randomization group) | 0 | 0
Cross Over at Week 24 | 60 (Study discontinuation/completion reported under randomization group) | 0 | 0
Qualified Re-randomization at Week 52 | 0 | 3 | 2
Completed | 0 | 0 | 0
Not Completed | 116 | 118 | 122
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lack of Efficacy | 6 | 6 | 4
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 4
Not completed — Study Terminated by Sponsor | 77 | 80 | 86
Not completed — Subject Refused Further Study Treatment | 0 | 1 | 0
Not completed — Other | 29 | 27 | 25

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all participants who were randomized and received at least one administration of study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg | Total
Number analyzed (Participants) | 116 | 118 | 122 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.75) | 33.9 (8.39) | 34.9 (9.06) | 34.3 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 65 | 59 | 176
  Male | 64 | 53 | 63 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 13 | 37
  Not Hispanic or Latino | 105 | 104 | 109 | 318
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 10 | 13 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 98 | 99 | 104 | 301
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 5 | 6 | 5 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 10 | 13 | 35
  Black or African American | 0 | 3 | 0 | 3
  Other | 10 | 14 | 12 | 36
  White Non-Hispanic | 94 | 91 | 97 | 282
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 0 | 4 | 6
  AUSTRALIA | 8 | 8 | 6 | 22
  BELGIUM | 8 | 10 | 9 | 27
  CZECH REPUBLIC | 11 | 8 | 8 | 27
  FRANCE | 6 | 5 | 3 | 14
  GERMANY | 2 | 9 | 7 | 18
  HUNGARY | 1 | 5 | 4 | 10
  MEXICO | 8 | 9 | 7 | 24
  POLAND | 18 | 11 | 16 | 45
  RUSSIAN FEDERATION | 18 | 22 | 22 | 62
  SOUTH KOREA | 6 | 1 | 5 | 12
  TAIWAN | 6 | 9 | 8 | 23
  UKRAINE | 18 | 19 | 20 | 57
  UNITED KINGDOM | 4 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 20 Response at Week 24
Description: ASAS 20 defined as improvement of greater than or equal to (>=) 20 % from baseline and absolute improvement from baseline of 1 on a 0 to 10 centimeter(cm) scale in at least 3 of following 4 domains: Patient's global assessment of disease activity (0 to 10 cm; 0=very well,10=very poor), total back pain (0 to 10 cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 to participant's ability to cope with everyday life), Inflammation (0 to 10 cm;0=none,10=very severe); absence of deterioration (>= 20% and worsening of at least 1 on a 0 to 10 cm scale) from baseline in remaining domain. ASAS20 response based on imputed data using treatment failure (consider non-responders at and after treatment failure),early escape rules (consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: Modified Full Analysis Set (MFAS)-participants who were randomized (those participants who would have been able to complete Week 24 at time of study discontinuation) and received at least 1 dose of study drug. Participants were analyzed per assigned treatment regardless of actual treatment received.
Measure: Number; unit: Percentage of participants
Groups:
- Ustekinumab 45 mg: Participants received ustekinumab 45 mg SC at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind.
- Ustekinumab 90 mg: Participants received ustekinumab 90 mg SC at Weeks 0 and 4, followed by every four weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind.
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants | 47.6 | 55.4 | 49.4

2. Secondary Outcome: Percentage of Participants Who Achieved an ASAS 40 Response at Week 24
Description: ASAS 40 defined as improvement of >= 40% from baseline and absolute improvement from baseline of at least 2 on 0 to 10 cm scale in at least 3 of following 4 domains: Patient's global assessment of disease activity (0 to 10 cm; 0=very well,10=very poor),total back pain (0 to 10 cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10 cm; 0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: MFAS- participants who were randomized (those participants who would have been able to complete Week 24 at time of study discontinuation) and received at least 1 dose of study drug. Participants were analyzed per assigned treatment regardless of actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants | 25.6 | 33.7 | 28.2

3. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Improvement From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24
Description: The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10 centimeter (cm) visual analog scale (VAS), with 0 being none, and 10 being very severe. In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness were added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom. 50% improvement in response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants | 23.2 | 32.5 | 25.9

4. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 24
Description: The BASFI is composed with 10 questions (each question is answered with a visual analogue scale 0-10 cm) to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of ankylosing spondylitis participants. Each question is a 10cm VAS with a value between 0 (easy) and 10 (impossible). The final BASFI score is the mean of the 10 scores. The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10. Higher BASFI score indicates more severe functional limitations of the participant due to AS. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 24
Population: MFAS population was included. Participants were analyzed per assigned treatment regardless of actual treatment received. 'N' (number of participants analyzed) signifies number of participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 61 | 72 | 63
Units on a scale | -2.11 (2.371) | -2.28 (2.625) | -1.90 (2.731)

5. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-reactive Protein (CRP) Inactive Disease (<1.3) at Week 24
Description: ASDAS includes CRP milligram per liter (mg/L); four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included total back pain(TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment(PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain)+ (0.110*PGA)+ (0.073*peripheral pain/swelling)+ (0.058* DMS)+ (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants | 7.3 | 14.5 | 12.9

6. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) Levels Through Week 24
Description: Change from baseline in hsCRP levels was reported. hsCRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing). Here 'n' signifies the number of participants who were analyzed at each specified timepoints, for each arm, respectively.
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: MFAS-participants who were randomized (those participants who would have been able to complete Week 24 at time of study discontinuation) and received at least 1 dose of study drug. Participants were analyzed per assigned treatment regardless of actual treatment received.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Milligrams per deciliter (mg/dL)
  Change at Week 4: number analyzed (Participants) | 82 | 83 | 84
  Change at Week 4 | -0.08 (1.567) | -0.10 (2.574) | -0.39 (1.601)
  Change at Week 8: number analyzed (Participants) | 82 | 82 | 82
  Change at Week 8 | -0.23 (1.490) | -0.53 (2.084) | -0.57 (2.209)
  Change at Week 12: number analyzed (Participants) | 80 | 81 | 81
  Change at Week 12 | -0.23 (1.661) | -0.71 (2.392) | -0.61 (2.534)
  Change at Week 16: number analyzed (Participants) | 79 | 82 | 80
  Change at Week 16 | -0.49 (1.725) | -0.63 (2.211) | -0.61 (2.539)
  Change at Week 20: number analyzed (Participants) | 61 | 80 | 80
  Change at Week 20 | -0.36 (1.951) | -0.78 (2.353) | -0.76 (2.383)
  Change at Week 24: number analyzed (Participants) | 62 | 79 | 79
  Change at Week 24 | -0.42 (2.145) | -0.63 (2.402) | -0.78 (2.413)

7. Secondary Outcome: Percentage of Participants With ASAS 20 Components at Week 24
Description: ASAS 20 defined as >= 20% improvement from baseline in 4 individual components of ASAS20: Patient's global assessment (PGA) of disease activity (0 to 10cm; 0=very well,10=very poor), total back pain(0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean(0 to10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to functional anatomy and 2 relate to participant's ability to cope with life) and Inflammation (0 to 10cm;0=none,10=very severe).
Time Frame: Week 24
Population: MFAS- participants who were randomized (those participants who would have been able to complete Week 24 at time of study discontinuation) and received at least 1 dose of study drug. Participants were analyzed per assigned treatment regardless of actual treatment received. 'N' signifies number of participants who were evaluable for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 78 | 80 | 80
Percentage of participants
  >=20% improvement from baseline in PGA score | 64.1 | 61.3 | 58.8
  >=20% improvement from baseline in total back pain | 62.8 | 60.0 | 60.0
  >=20% improvement from baseline in BASFI | 53.8 | 57.5 | 56.3
  >=20% improvement from baseline in inflammation | 64.1 | 66.3 | 65.0

8. Secondary Outcome: Percentage of Participants Who Achieved ASAS 40 Response at Week 4, 8, 12, 16 and 20
Description: ASAS 40 defined as improvement of >= 40% from baseline and absolute improvement from baseline of at least 2 on 0 to10cm scale in at least 3 of following 4 domains: Patient's global assessment of disease activity (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure (consider non-responders at and after treatment failure), early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants
  Week 4 | 3.7 | 8.4 | 11.8
  Week 8 | 18.3 | 19.3 | 18.8
  Week 12 | 17.1 | 27.7 | 24.7
  Week 16 | 19.5 | 27.7 | 24.7
  Week 20 | 24.4 | 38.6 | 32.9

9. Secondary Outcome: Percentage of Participants Who Achieved ASAS 20 Response at Week 4, 8, 12, 16 and 20
Description: ASAS 20 defined as improvement of >= 20 % from baseline and absolute improvement from baseline of 1 on a 0 to 10 cm scale in at least 3 of following 4 domains: Patient's global assessment of disease activity (0 to 10 cm; 0=very well,10=very poor), total back pain (0 to 10 cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 to participant's ability to cope with everyday life), Inflammation (0 to 10 cm;0=none,10=very severe); absence of deterioration (>= 20% and worsening of at least 1 on a 0 to 10 cm scale) from baseline in remaining domain. ASAS20 response based on imputed data using treatment failure (consider non-responders at and after treatment failure),early escape rules (consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants
  Week 4 | 23.2 | 26.5 | 32.9
  Week 8 | 31.7 | 41.0 | 36.5
  Week 12 | 34.1 | 48.2 | 41.2
  Week 16 | 40.2 | 49.4 | 35.3
  Week 20 | 45.1 | 59.0 | 44.7

10. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Improvement From Baseline in BASDAI at Week 4, 8, 12, 16 and 20
Description: The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10 centimeter (cm) visual analog scale (VAS), with 0 being none, and 10 being very severe. In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness will be added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom. 50% improvement in BASDAI based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non-responders).
Time Frame: Week 4, 8, 12, 16, and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants
  Week 4 | 4.9 | 8.4 | 8.2
  Week 8 | 9.8 | 15.7 | 17.6
  Week 12 | 18.3 | 16.9 | 28.2
  Week 16 | 19.5 | 21.7 | 24.7
  Week 20 | 15.9 | 28.9 | 32.9

11. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 4, 8, 12, 16 and 20
Description: The BASFI is composed with 10 questions (each question is answered with a visual analogue scale 0-10 cm) to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Each question is a 10cm VAS with a value between 0 (easy) and 10 (impossible). The final BASFI score is the mean of the 10 scores. The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10. Higher BASFI score indicates more severe functional limitations of the participant due to AS. Missing data were imputed using early escape rule (measurement value at Week 20 and 24 was set as missing). Here 'n' defined as number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Time Frame: Baseline, Week 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Units on a scale
  Change at Week 4: number analyzed (Participants) | 82 | 83 | 84
  Change at Week 4 | -0.60 (1.582) | -1.15 (1.748) | -0.79 (1.600)
  Change at Week 8: number analyzed (Participants) | 82 | 82 | 82
  Change at Week 8 | -0.82 (1.997) | -1.54 (2.177) | -1.05 (2.095)
  Change at Week 12: number analyzed (Participants) | 79 | 82 | 80
  Change at Week 12 | -1.00 (2.064) | -1.69 (2.079) | -1.35 (2.458)
  Change at Week 16: number analyzed (Participants) | 81 | 82 | 80
  Change at Week 16 | -1.05 (2.162) | -1.75 (2.312) | -1.17 (2.747)
  Change at Week 20: number analyzed (Participants) | 61 | 80 | 80
  Change at Week 20 | -1.70 (2.339) | -2.11 (2.394) | -1.64 (2.794)

12. Secondary Outcome: Percentage of Participants With ASDAS (CRP) Inactive Disease (<1.3) at Week 4, 8, 12, 16, and 20
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included total back pain(TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment(PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain)+ (0.110*PGA)+ (0.073*peripheral pain/swelling)+ (0.058* DMS)+ (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16, and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 82 | 83 | 85
Percentage of participants
  Week 4 | 2.4 | 3.6 | 1.2
  Week 8 | 6.1 | 7.2 | 9.4
  Week 12 | 4.9 | 4.8 | 10.6
  Week 16 | 6.1 | 7.2 | 11.8
  Week 20 | 3.7 | 13.3 | 15.3

ADVERSE EVENTS:
Time Frame: Approximately up to 2.2 years
Description: The safety analysis set included all participants who received at least 1 (partial or complete) administration of study agent, i.e., the treated population. In the safety analyses, participants were analyzed according to the treatment they actually received, regardless of their randomized treatments.
Groups:
- Placebo Only: Participants received placebo SC at Week 0, 4, 16 and 20. At Week 16, participants in placebo group who qualified for EE criteria (with <10 % improvement from baseline in both total back pain and morning stiffness measures at Week 12 and 16) re-randomized to receive ustekinumab 45mg or 90mg at Week 16, 20 and 28 followed by q12w dosing through Week 52. Participants received placebo SC at Week 24 to maintain the blind. At Week 24, remaining participants in placebo group who did not meet EE criteria were re-randomized to receive ustekinumab 45mg or 90mg at Week 24 and 28 followed by q12w therapy through Week 52. At Week 52, participants who achieved inactive disease [ASDAS] [ESR]<1.3 at both Week 40 and 52 underwent re-randomization to either Ustekinumab or placebo. Participants who did not achieve inactive disease at either Week 40 or 52 received previously assigned Ustekinumab dose at scheduled visits.
- Placebo to Ustekinumab 45mg: Participants randomized to placebo SC at Week 0 and re-randomized to early escape at Week 16 or cross over at Week 24 to ustekinumab 45 mg SC; adverse events are counted from crossover onward. All participants regardless qualified for re-randomization at Week 52 or not were counted.
- Placebo to Ustekinumab 90mg: Participants randomized to placebo SC at week 0 and re-randomized to early escape at Week 16 or cross over at Week 24 to ustekinumab 90 mg SC; adverse events are counted from crossover onward. All participants regardless qualified for re-randomization at Week 52 or not were counted.
- Ustekinumab 45mg Only: Participants received ustekinumab 45 mg subcutaneously (SC) at Weeks 0 and 4, followed by every 12 weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind. At Week 52, all participants who achieved inactive disease (ASDAS ESR<1.3) at both Week 40 and 52 underwent re-randomization to either remain on ustekinumab or placebo. Participants who did not achieve inactive disease at either Week 40 or 52 received previously assigned ustekinumab dose at their scheduled visits. All participants regardless qualified for re-randomization at Week 52 or not were counted.
- Ustekinumab 90mg Only: Participants received ustekinumab 90 mg subcutaneously at Weeks 0 and 4, followed by every four weeks through Week 52. At Weeks 20 and 24, participants received placebo subcutaneously to maintain the blind.At Week 52, all participants who achieved inactive disease (ASDAS ESR<1.3) at both Week 40 and 52 underwent re-randomization to either remain on ustekinumab or placebo. Participants who did not achieve inactive disease at either Week 40 or 52 received previously assigned ustekinumab dose at their scheduled visits. All participants regardless qualified for re-randomization at Week 52 or not were counted.
Arm/Group | Placebo Only | Placebo to Ustekinumab 45mg | Placebo to Ustekinumab 90mg | Ustekinumab 45mg Only | Ustekinumab 90mg Only
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/42 | 0/40 | 0/118 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/116 | 0/42 | 2/40 | 2/118 | 6/122
Other Adverse Events (participants affected / at risk) | 19/116 | 4/42 | 12/40 | 27/118 | 27/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Only (N=116) | Placebo to Ustekinumab 45mg (N=42) | Placebo to Ustekinumab 90mg (N=40) | Ustekinumab 45mg Only (N=118) | Ustekinumab 90mg Only (N=122)
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Axial Spondyloarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Only (N=116) | Placebo to Ustekinumab 45mg (N=42) | Placebo to Ustekinumab 90mg (N=40) | Ustekinumab 45mg Only (N=118) | Ustekinumab 90mg Only (N=122)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 2
Fatigue (General disorders) | 2 | 0 | 4 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 2 | 5 | 8
Viral Upper Respiratory Tract Infection (Infections and infestations) | 6 | 1 | 1 | 11 | 9
Alanine Aminotransferase Increased (Investigations) | 3 | 1 | 2 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 2 | 3
Headache (Nervous system disorders) | 1 | 0 | 2 | 3 | 4

LIMITATIONS AND CAVEATS:
The study was discontinued before it was fully enrolled, therefore, the interpretation of the efficacy data is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2015-04-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT02407223/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT02407223/SAP_001.pdf